CLINICAL TRIAL: NCT04786262
Title: A Phase 1/2/3 Study to Evaluate the Safety, Tolerability, and Efficacy of VX-880 in Subjects Who Have Type 1 Diabetes Mellitus With Impaired Hypoglycemic Awareness and Severe Hypoglycemia
Brief Title: A Safety, Tolerability, and Efficacy Study of VX-880 in Participants With Type 1 Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX20-880-101; 2024-513929-23-00 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 1; Impaired Hypoglycemic Awareness; Severe Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-880 (Experimental)
  Interventions: Biological: VX-880

INTERVENTIONS:
Biological: VX-880 — Infused into the hepatic portal vein.
  Other Names: Zimislecel; Formerly known as STx-02

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of VX-880 infusion in participants with Type 1 diabetes (T1D) and impaired awareness of hypoglycemia (IAH) and severe hypoglycemia.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical history of T1D with > 5 years of duration of insulin dependence
* At least two episodes of documented severe hypoglycemia in the 12 months prior to enrollment
* Stable diabetic treatment
* Consistent use of continuous glucose monitor (CGM) for at least 3 months before Screening and willingness to use CGM for the duration of the study

Key Exclusion Criteria:

-Prior islet cell transplant, organ transplant, or cell therapy

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) | From VX-880 infusion to end of study (up to 5 years)
Parts B and C: Proportion of Participants who are Insulin Independent with Absence of Severe Hypoglycemic Events (SHEs) | 1 year after achieving insulin independence

SECONDARY OUTCOMES:
Parts B and C: Proportion of Participants who are Insulin Independent | At 1 year after VX-880 infusion
Parts B and C: Proportion of Participants Free from SHEs with a Glycosylated Hemoglobin (HbA1c) less than (<) 7.0% | At 1 year after VX-880 infusion
Parts B and C: Change From Baseline in Glycosylated Hemoglobin (HbA1c) | At 1 year after VX-880 infusion
Parts B and C: Proportion of Participants Who Maintain Insulin Independence for at least 1 year | From VX-880 infusion to end of study (up to 5 years)
Parts B and C: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) | From Signing of informed consent to end of study (up to 5 years)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (12):
  - City of Hope, Duarte, California
  - University of California San Francisco, San Francisco, California
  - UHealth Diabetes Research Institute, Miami, Florida
  - Northwestern Organ Transplant Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Montefiore, Pittsburgh, Pennsylvania
  - Baylor Scott and White Research Institute, Dallas, Texas
  - VCU Medical Center, Richmond, Richmond, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Canada (4):
  - University of Alberta, Edmonton, Edmonton
  - McGill University Health Centre, Montreal
  - Toronto General Hospital (TGH), Toronto
  - Vancouver General Hospital, Vancouver
- France (2):
  - CHU Lille, Lille
  - Centre de recherche en Biomédecine de Strasbourg, Strasbourg
- Dresden Center for Islet Transplantation, Dresden, Germany
- IRCCS Ospedale San Raffaele, Milan, Italy
- Leiden University, Leiden, Netherlands
- Oslo University Hospital, Oslo, Norway
- Saudi Arabia (2):
  - King Abdullah International Medical Research Center (KAIMRC) - Riyadh - Endocrinology, Riyadh
  - King Faisal Specialist Hospital & Research Centre - Riyadh - Endocrinology, Riyadh
- Hopiteaux Universitaires de Geneve, Geneva, Switzerland
- United Kingdom (4):
  - Churchill Hospital, Headington, Oxford
  - Royal Infirmary of Edinburgh, Edinburgh
  - Cardiovascular, Metabolic Medicine and Sciences, King's College London, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Reichman TW, Markmann JF, Odorico J, Witkowski P, Fung JJ, Wijkstrom M, Kandeel F, de Koning EJP, Peters AL, Mathieu C, Kean LS, Bruinsma BG, Wang C, Mascia M, Sanna B, Marigowda G, Pagliuca F, Melton D, Ricordi C, Rickels MR; VX-880-101 FORWARD Study Group. Stem Cell-Derived, Fully Differentiated Islets for Type 1 Diabetes. N Engl J Med. 2025 Sep 4;393(9):858-868. doi: 10.1056/NEJMoa2506549. Epub 2025 Jun 20. PMID 40544428